CLINICAL TRIAL: NCT06227637
Title: Local Muscle Vibration Versus Muscle Energy Technique In Sacroiliac Joint Dysfunction
Acronym: SIJD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Abou Almakarem Ali Radwan, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: local vibration vs MET in SIJD
Record Dates: First submitted 2024-01-11; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Intervention Model Description: The sample will be randomly subdivided into 2 Groups: Group (A)- Muscle Energy Techniques and Group (B)- Local Muscle Vibration.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to the treatment they will receive, and the statistics doctor will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Muscle Energy Techniques ) (Active Comparator): Muscle Energy Techniques
  Interventions: Other: Local Muscle Vibration compared to Muscle energy technique in SIJD
- Group( B) (Local Muscle Vibration) (Active Comparator): Local Muscle Vibration
  Interventions: Other: Local Muscle Vibration compared to Muscle energy technique in SIJD

INTERVENTIONS:
Other: Local Muscle Vibration compared to Muscle energy technique in SIJD — Apply Local Muscle Vibration compared to Muscle energy technique on patients with sacroiliac joint dysfunction and note the effect on pain intensity, pain pressure threshold, functional disability, and innominate angle tilt in SIJD.

SUMMARY:
The purpose of this study is to compare the effect of Local Muscle Vibration versus Muscle energy technique on pain intensity, pain pressure threshold, functional disability, and innominate angle tilt in SIJD.

This study will try to answer the following question:

What is the effect of Local Muscle Vibration compared to Muscle energy technique on pain intensity, pain pressure threshold, functional disability, and innominate angle tilt in SIJD?

DETAILED DESCRIPTION:
Clinicians will attempt to identify the primary factors that contribute to the development of low back pain. These factors are related to specific areas of malfunction that may irritate the tissues and create pain, or cause pain through hypersensitivity of nociceptive pathways in the CNS. Joint dysfunction is one risk factor, which is defined as "loss of joint play movement that cannot be produced by voluntary muscles". Pain in the joint can result from joint dysfunction, in addition to joint dysfunction, muscle dysfunction is evaluated. History, inspection, palpation, and flexibility tests can all be used to determine this.

Muscle energy technique is based on the concepts of Autogenic Inhibition and Reciprocal Inhibition, to lengthen a shortened muscle, mobilize a stiff joint, strengthen a weak muscle, and reduce localized edema and passive congestion. Several studies approved that (MET) affects positively on SIJD cases.

Local Muscle Vibration is used to pain relief, stimulate edema absorption, improve blood flow, alleviate wound healing, and for its anti-inflammatory and ant-adhesion effects. In addition, pain relief effect have also been widely demonstrated. Vibration comprised of low-magnitude high-intensity stimuli which represents a suitable technique to securely transmit appropriate mechanical signals to patients who are unable to exercise to increase musculoskeletal strength. According to a narrative literature review contain about 35 study descuss effects of local vibration therapy on various performance parameters, LMV have apositive effect on muscle activation, strengh, power and joint range of motion.

According to Iodice et al (2011), local administration of high-frequency VT resulted in significant increase in muscle function after several weeks however, some hormonal alterations and moderate performance gains were observed after a single session. This study will try to investigate the effect of Local Muscle Vibration versus Muscle energy technique, which is more effective in reducing low back pain and disability in cases of SIJD. Up to the authors knowledge no previous study discussed the difference between (LMV) and (MET) on SIJD.

ELIGIBILITY:
Inclusion Criteria:

both male and female participants with ages between 20-40.

* Pain intensity is greater than 3 over the scale of VAS.
* Pain around SIJ (around PSIS and sacral sulcus).
* Participants with at least three positives out of six provocation and motion palpation tests that have been validated (distraction, compression, Gaenslen, posterior friction test, sacral thrust, and FABER tests).

Exclusion Criteria:

* Neurological impairments in the leg
* Sacroiliitis
* Spondylolisthesis
* pre-diagnosed central or peripheral nervous system disease
* The current pregnancy
* rheumatoid arthritis
* Major surgery of lower limbs and spine

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Assessment before treatment, then immediately after the intervention, then finally follow up after 2 weeks
  VAS in the simple model, which will be used as a self-reported method of pain intensity measurement, the patient will be asked to put a mark point at the scale range (from 0 to 10 cm). This assessment procedure will be applied before and after treatment procedure.
Pain pressure threshold | Assessment before treatment, then immediately after the intervention, then finally follow up after 2 weeks
  PPT should be measured on both sides at the level of right and left posterior inferior iliac spines (PIIS). With the patient is a prone position, two algometer measurements will be taken before and after treatment at the level of (PIIS). All measurements will be recorded at intervals of 30 second. The patient will be instructed to report when the sensation beginning of pain.
Back functional disability | Assessment before treatment, then immediately after the intervention, then finally follow up after 2 weeks
  This questionnaire is Self-reported pain and disability method (Arabic model). The therapist will ask the patient ten questions covering pain severity, personal care, lifting, walking, sitting, standing, sleeping, social life, travelling, and changing degrees of pain. Each part has six statements, each with a score ranging from 0 (showing no disability) to 5 (representing maximum disability). The final score was calculated as a percentage out of 50, representing perceived disability at the time. The validated Arabic version of ODI will be used in this study.
The innominate angle tilt | Assessment before treatment, then immediately after the intervention, then finally follow up after 2 weeks
  The patient will be instructed to march 10 steps in place before standing in a fully erect posture without bending ankles, knees, or hips, feet in front 30.5 cm apart, and arms across the chest. The therapist will stand beside the patient and mark the anterior and posterior superior iliac spines (ASIS and PSIS).

CONTACTS AND LOCATIONS:
Overall Officials: Mona M ibrahim, Doctorate, Study Chair — Cairo University; Enas F youssef, Doctorate, Study Chair — Cairo University
Locations (1):
- The faculty of physical therapy, Cairo university, and Gezira Youth Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Germann D, El Bouse A, Shnier J, Abdelkader N, Kazemi M. Effects of local vibration therapy on various performance parameters: a narrative literature review. J Can Chiropr Assoc. 2018 Dec;62(3):170-181. PMID 30662072
- [Background] Konrad A, Glashuttner C, Reiner MM, Bernsteiner D, Tilp M. The Acute Effects of a Percussive Massage Treatment with a Hypervolt Device on Plantar Flexor Muscles' Range of Motion and Performance. J Sports Sci Med. 2020 Nov 19;19(4):690-694. eCollection 2020 Dec. PMID 33239942
- See also: Alkady, S. M. E., Kamel, R. M., AbuTaleb, E., Lasheen, Y., & Alshaarawy, F. A. (2019). Effect of Muscle Energy Technique in Chronic Sacroiliac Joint Dysfunction. South Valley University International Journal of Physical Therapy and Sciences, 1(1), 8-19. — https://doi.org/10.21608/svupts.2019.230984
- See also: Salvador Coloma, P., & Sánchez-Zuriaga, D. (2019). Effects of myofascial release in erector spinae myoelectric activity and lumbar spine kinematics in non-specific chronic low back pain: Randomized controlled trial. Clinical Biomechanics, 63(1), 27-33. — https://doi.org/10.1016/j.clinbiomech.2019.02.009
- See also: Azevedo, D. C., Santos, H., Carneiro, R. L., & Andrade, G. T. (2014). Reliability of sagittal pelvic position assessments in standing, sitting and during hip flexion using palpation meter. Journal of Bodywork and Movement Therapies, 18(2), 210-214. — https://doi.org/10.1016/j.jbmt.2013.05.017
- See also: Posterior , Lateral , and Anterior Hip Pain Due to Musculoskeletal Origin : A Narrative Literature Review of History , Physical Examination , and Diagnostic Imaging. Journal of Chiropractic Medicine, 15(4), 281-293. — https://doi.org/10.1016/j.jcm.2016.08.004
- See also: Chan, M. E., Uzer, G., & Rubin, C. T. (2013). The potential benefits and inherent risks of vibration as a non-drug therapy for the prevention and treatment of osteoporosis. Current Osteoporosis Reports, 11(1), 36-44. — https://doi.org/10.1007/s11914-012-0132-1
- See also: Cohen, S. P. (2005). Sacroiliac Joint Pain : A Comprehensive Review of Anatomy , Diagnosis , and Treatment. Anesthesia & Analgesia, 101(5), 1440-1453. — https://doi.org/10.1213/01.ANE.0000180831.60169.EA
- See also: De Gail, P., Lance, J. W., & Neilson, P. D. (1966). Differential effects on tonic and phasic reflex mechanisms produced by vibration of muscles in man. Journal of Neurology, Neurosurgery, and Psychiatry, 29(1), 1-11. — https://doi.org/10.1136/jnnp.29.1.1
- See also: Dueñas, L., Zamora, T., Lluch, E., Artacho-Ramírez, M. A., Mayoral, O., Balasch, S., & Balasch-Bernat, M. (2020). The effect of vibration therapy on neck myofascial trigger points: A randomized controlled pilot study. Clinical Biomechanics, 78(May 2019), — https://doi.org/10.1016/j.clinbiomech.2020.105071
- See also: Increase in paravertebral muscle activity in lumbar kyphosis patients by surface electromyography compared with lumbar spinal canal stenosis patients and healthy volunteers. The Spine Journal, 13(11), 1711. — https://doi.org/10.1016/j.spinee.2013.10.009
- See also: Feeney, D. F., Capobianco, R. A., Montgomery, J. R., Morreale, J., Grabowski, A. M., & Enoka, R. M. (2018). Individuals with sacroiliac joint dysfunction display asymmetrical gait and a depressed synergy between muscles providing sacroiliac joint force — https://doi.org/10.1016/j.jelekin.2018.09.009
- See also: Fritton, S. P., J. McLeod, K., & Rubin, C. T. (2000). Quantifying the strain history of bone: Spatial uniformity and self-similarity of low-magnitude strains. Journal of Biomechanics, 33(3), 317-325. — https://doi.org/10.1016/S0021-9290(99)00210-9
- See also: Fryer, G., & Pearce, A. J. (2013). The effect of muscle energy technique on corticospinal and spinal reflex excitability in asymptomatic participants. Journal of Bodywork and Movement Therapies, 17(4), 440-447. — https://doi.org/10.1016/j.jbmt.2013.05.006
- See also: Gartenberg, A., Nessim, A., & Cho, W. (2021). Sacroiliac joint dysfunction : pathophysiology , diagnosis , and treatment. European Spine Journal, 30(10), 2936-2943. — https://doi.org/10.1007/s00586-021-06927-9
- See also: Goebel, R. T., Kleinöder, H., Yue, Z., Gosh, R., & Mester, J. (2015). Effect of Segment-Body Vibration on Strength Parameters. Sports medicine - open, 1(1), 14. — https://doi.org/10.1186/s40798-015-0022-z
- See also: Harkins&, I, D. D. P., Bush, F. M., Long, S., S. W. (1993). A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain, 56(2), 21-226. — https://doi.org/10.1016/0304-3959(94)90097-3
- See also: Henricson, A., Larsson, A., Olsson, E., & Westlin, N. (1983). The effect of stretching on the range of motion of the ankle joint in badminton players. Journal of Orthopaedic and Sports Physical Therapy, 5(2), 74-77. — https://doi.org/10.2519/jospt.1983.5.2.74
- See also: Holey, L. (1996). Muscle Energy Techniques. Physiotherapy, 82(8), 493. — https://doi.org/10.1016/s0031-9406(05)66417-6
- See also: Hussein, Y. I., Hassan, K. A., & EL-Nahass, B. G. E. (2022). Strain-counterstrain versus muscle energy technique in sacroiliac joint dysfunction. International Journal of Health Sciences, 6(July), 8738-8754. — https://doi.org/10.53730/ijhs.v6ns4.10935
- See also: Iodice, P., Bellomo, R. G., Gialluca, G., Fanò, G., & Saggini, R. (2011). Acute and cumulative effects of focused high-frequency vibrations on the endocrine system and muscle strength. European Journal of Applied Physiology, 111(6), 897-904. — https://doi.org/10.1007/s00421-010-1677-2
- See also: Ivanov, A. A., Kiapour, A., Ebraheim, N. A., & Goel, V. (2009). Lumbar Fusion Leads to Increases in Angular Motion and Stress Across Sacroiliac Joint A Finite Element Study. Spine, 34(5), 162-169. — https://doi.org/10.1097/BRS.0b013e3181978ea3
- See also: Kiapour, A. L. I., Joukar, A., Elgafy, H., & Erbulut, D. U. (2020). Biomechanics of the Sacroiliac Joint : Anatomy , Function , Biomechanics , Sexual Dimorphism , and Causes of Pain. Journal of Pain Research, 14(1), 3135-3143. — https://doi.org/10.2147/JPR.S327351
- See also: Diagnosing painful sacroiliac joints : A validity study of a McKenzie evaluation and sacroiliac provocation tests. Australian Journal of Physiotherapy, 49(2), 89-97. — https://doi.org/10.1016/S0004-9514(14)60125-2
- See also: The acute effects of local muscle vibration frequency on peak torque, rate of torque development, and EMG activity. Official Journal of the International Society of Electrophysiological Kinesiology. 24(6), 888-894. — https://doi.org/10.1016/j.jelekin.2014.07.014
- See also: "Effectiveness of Manipulation and Muscle Energy Techniques in Subjects with SI Joint Dysfunction." nternational Journal of Pharmaceutical Science and Health Care 4(5): 16-29. — https://www.researchgate.net/publication/281775681
- See also: Effects of local vibrations on skeletal muscle trophism in elderly people: mechanical, cellular, and molecular events. International journal of molecular medicine, 24(4), 503-512. — https://doi.org/10.3892/ijmm_00000259
- See also: Deformation of the innominate bone and mobility of the pubic symphysis during asymmetric moment application to the pelvis. Manual Therapy, 17(1), 66-70. — https://doi.org/10.1016/j.math.2011.09.002
- See also: Prather, H., Bonnette, M., & Hunt, D. (2020). Nonoperative Treatment Options for Patients With Sacroiliac Joint Pain. International Journal of Spine Surgery, 14, 35-40. — https://doi.org/10.14444/6082
- See also: Prather, H., & Hunt, D. (2004). Sacroiliac Joint Pain. Disease-a-Month, 50(12), 670-683. — https://doi.org/10.1016/j.disamonth.2004.12.004
- See also: Ramzy, R. (2008). Validation of the Arabic Version of the Oswestry Disability Index Developed in Tunisia for low back pain patients in the UAE. — https://core.ac.uk/download/pdf/37321542.pdf
- See also: Effects of Muscle Energy Technique versus Mobilization on Pain and Disability in Post-Partum Females with Sacroiliac Joint Dysfunction. In Indian Journal of Health Sciences and Care, 5(1), 11. — https://doi.org/10.5958/2394-2800.2018.00003.2
- See also: A randomized clinical trial of manual versus mechanical force manipulation in the treatment of sacroiliac joint syndrome. Journal of Manipulative and Physiological Therapeutics, 28(7), 493-501. — https://doi.org/10.1016/j.jmpt.2005.07.006
- See also: Effect of Sacroiliac Joint Mobilization on the Level of Soft Tissue Pain Threshold in Asymptomatic Women. Journal of Manipulative and Physiological Therapeutics, 41(3), 258-264. — https://doi.org/10.1016/j.jmpt.2017.09.004
- See also: New concepts and hypotheses Transfer of lumbosacral load to iliac bones and legs Part 1 : Biomechanics of self-bracing of the sacroiliac joints and its significance for treatment and exercise. Clinical Biomechanics, 8(6), 285-294. — https://doi.org/10.1016/0268-0033(93)90002-Y
- See also: Szadek, K. M., Wurff, P. Van Der, Tulder, M. W. Van, Zuurmond, W. W., & Perez, R. S. G. M. (2009). Diagnostic Validity of Criteria for Sacroiliac Joint Pain : The Journal of Pain, 10(4), 354-368. — https://doi.org/10.1016/j.jpain.2008.09.014
- See also: Effect of the single-leg, lateral oblique, decline squat exercise on sacroiliac joint pain with knee pain. Journal of Physical Therapy Science, 28(9), 2688-2689. — https://doi.org/10.1589/jpts.28.2688
- See also: Zunzunwala, S., Phansopkar, P., & Lakhwani, M. (2022). Effect of theragun on calf muscle tightness in asymptomatic individuals. Journal of Medical Pharmaceutical and Allied Sciences, 11(3), 4863-4866. — https://doi.org/10.55522/jmpas.V11I3.1364